CLINICAL TRIAL: NCT03352531
Title: A Phase 1A/1B Multicenter, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK105 in Subjects With Advanced Solid Tumors
Brief Title: Study of the Safety, Pharmacokinetics, and Antitumor Activity of AK105 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK105-101
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced Cancer
Keywords: Anti-PD-1 monoclonal antibody; immunotherapy; immuno-oncology; advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK-105 (Experimental): Single-arm
  Interventions: Biological: AK-105

INTERVENTIONS:
Biological: AK-105 — Anti-PD-1 monoclonal antibody; Subjects will receive AK105 by intravenous administration.

SUMMARY:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of AK105 as a single agent in adult subjects with advanced solid tumor malignancies. The study consists of a dose escalation phase (Phase 1a) to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for AK105 as a single agent, and a dose expansion phase (Phase 1b) in subjects with specific tumor types which will characterize treatment of AK105 as a single agent at the MTD or RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent and any locally required authorization obtained from the subject/legal representative.
* In dose-escalation cohorts (Phase 1a), histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.
* In the dose-expansion cohorts (Phase 1b), histologically or cytologically confirmed selected advanced solid tumors.
* Subject must have at least one measurable lesion according to RECIST Version1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.
* Available archived tumor tissue sample to allow for correlative biomarker studies. In the setting where archival material is unavailable or unsuitable for use, the subject must consent and undergo fresh tumor biopsy.
* Adequate organ function.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs.
* For dose-escalation phase (Phase 1a), prior exposure to any anti-PD-1, anti-PD-L1, anti-CTL4 antibody. For dose-expansion phase (Phase 1b), prior exposure to any anti-PD-1, anti-PD-L1, anti-CTL4 antibody or any other antibody or drug targeting T-cell costimulation or checkpoint pathways such as ICOS, or agonists such as CD40, CD137, GITR, OX40 etc.
* Receipt of any immunotherapy, any conventional or investigational systemic anticancer therapy within 4 weeks prior to the first dose of AK105.
* Prior treatment with systemic immune modulating agents (other than agents specified above) that was within 28 days prior to enrollment, or within 90 days prior to enrollment if there was an immune related adverse event, or associated with toxicity that resulted in discontinuation of the immune modulating agent.
* Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer related conditions is acceptable.
* Subjects with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
* Active or prior documented autoimmune disease within the past 2 years.
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency.
* History of organ transplant or hematopoietic stem cell that requires use of immunosuppressives.
* Known allergy or reaction to any component of the AK105 formulation.
* History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
* Known history of tuberculosis.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Known active hepatitis B or C infections, or any positive test at screening for hepatitis B or C virus indicating acute or chronic infection except for subjects with HCC. Subjects with past or resolved HBV infection are eligible. Subjects positive for HCV antibody are eligible only if qualitative HCV RNA tests is negative.
* An active infection requiring systemic therapy with the exception of antiviral therapy for hepatitis as specified by the protocol.
* Receipt of live or attenuated vaccination within 30 days prior to the first dose of AK105.
* Active or prior documented esophageal or gastric variceal bleeding
* Clinically apparent ascites on physical examination. Ascites that requires active ongoing paracentesis (within 6 weeks prior to the first scheduled dose) to control symptoms. Note: ascites detectable on imaging studies only are allowed.
* Portal vein invasion at the main portal (Vp4), inferior vena cava, or cardiac involvement of HCC based on imaging.
* Clinically diagnosed hepatic encephalopathy characterized by asterixis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the time of informed consent signed through 90 days after the last dose of AK105
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 4 weeks
  DLTs will be assessed during the first 4 weeks of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (4 weeks) of treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK105 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK105 until death due to any cause.
Area under the curve (AUC) of AK105 | From first dose of AK105 through 30 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Maximum observed concentration (Cmax) of AK105 | From first dose of AK105 through 30 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Minimum observed concentration (Cmin) of AK105 at steady state | From first dose of AK105 through 30 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through to 90 days after last dose of AK105
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - St Vincent's Hospital, Sydney (The Kinghorn Cancer Centre), Darlinghurst, New South Wales
  - Border Medical Oncology, East Albury, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - ICON Cancer Foundation, South Brisbane, Queensland
  - Ashford Cancer Centre Research, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Pang X, Zhong T, Qu T, Chen N, Ma S, He X, Xia D, Wang M, Xia M, Li B. Penpulimab, an Fc-Engineered IgG1 Anti-PD-1 Antibody, With Improved Efficacy and Low Incidence of Immune-Related Adverse Events. Front Immunol. 2022 Jun 27;13:924542. doi: 10.3389/fimmu.2022.924542. eCollection 2022. PMID 35833116
- [Derived] Zheng Y, Mislang ARA, Coward J, Cosman R, Cooper A, Underhill C, Zhu J, Xiong J, Jiang O, Wang H, Xie Y, Zhou Y, Jin X, Li B, Wang ZM, Kwek KY, Xia D, Xia Y, Xu N. Penpulimab, an anti-PD1 IgG1 antibody in the treatment of advanced or metastatic upper gastrointestinal cancers. Cancer Immunol Immunother. 2022 Oct;71(10):2371-2379. doi: 10.1007/s00262-022-03160-1. Epub 2022 Feb 15. PMID 35165764
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35165764/